CLINICAL TRIAL: NCT03320044
Title: Genetic Variations,Immuno-sequencing and Circulating Tumor DNA(ctDNA) for Early Diagnosis of Small Pulmonary Nodules
Brief Title: Early Diagnosis of Small Pulmonary Nodules by Multi-omics Sequencing
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1702
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Lung Neoplasm
Keywords: Circulating Tumor DNA; Lung cancer Surgery; early diagnosis; immuno-sequencing
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample from patient with small pulmonary nodule before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analyse immune repertoire and genetic mutations of benign and malignant pulmonary nodule，and evaluate peripheral blood detection for identifying nature of pulmonary nodule.

DETAILED DESCRIPTION:
Early diagnosis of lung cancer is of vital importance in lung cancer treatment. This research will first analyse the features of immune repertoire and genetic mutations from tissue of benign and malignant pulmonary nodule，then explore the feasibility of detecting these features from peripheral blood sample, and finally evaluate peripheral blood detection of lung cancer related immune repertoire and genetic mutations for identifying nature of pulmonary nodule.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent and consent to participate in this study;
2. Found small nodules in pulmonary by CT and prepare for surgery;

Exclusion Criteria:

1. Malignant tumor history within the past 5 years;
2. Receiving chemotherapy, radiotherapy or targeted therapy before surgery;
3. Histology confirmed not non-small cell lung cancer
4. No matching tissue or blood samplesUnqualified blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient are found small nodules in pulmonary and prepare for surgery
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of combining peripheral plasma circulating tumor DNA and white cell immuno-sequencing in diagnosis of early stage non-small cell lung cancer | 6 months

SECONDARY OUTCOMES:
The sensitivity and specificity of tissue immune repertoire in diagnosis of early stage non-small cell lung cancer | 6 months
The concordance of peripheral plasma circulating tumor DNA and tumor tissue DNA in diagnosis of early stage non-small cell lung cancer | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen K, Bai J, Reuben A, Zhao H, Kang G, Zhang C, Qi Q, Xu Y, Hubert S, Chang L, Guan Y, Feng L, Zhang K, Zhang K, Yi X, Xia X, Cheng S, Yang F, Zhang J, Wang J. Multiomics Analysis Reveals Distinct Immunogenomic Features of Lung Cancer with Ground-Glass Opacity. Am J Respir Crit Care Med. 2021 Nov 15;204(10):1180-1192. doi: 10.1164/rccm.202101-0119OC. PMID 34473939